CLINICAL TRIAL: NCT04121403
Title: Norwegian Study of Oral Cladribine and Rituximab in Multiple Sclerosis (NOR-MS) A Prospective Randomized Open-label Blinded Endpoint (PROBE) Multicenter Non-inferiority Study
Brief Title: Norwegian Study of Oral Cladribine and Rituximab in Multiple Sclerosis (NOR-MS)
Acronym: NOR-MS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Sykehuset Ostfold (Other); Sykehuset Telemark (Other Government); Vestre Viken Hospital Trust (Other); Sorlandet Hospital HF (Other Government); Helse Stavanger HF (Other Government); Sykehuset Innlandet HF (Other); Sykehuset i Vestfold HF (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Gro Owren Nygaard, Gro Owren Nygaard, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11383
Record Dates: First submitted 2019-09-23; First posted 2019-10-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Relapsing Multiple Sclerosis; Multiple Sclerosis
Keywords: multiple sclerosis; ms; rms; rituximab; cladribine; probe
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rituximab; Cladribine

STUDY DESIGN:
Intervention Model Description: A prospective randomized open-label blinded endpoint (PROBE) multicenter non-inferiority study, designed to establish non-inferiority of the test treatment rituximab compared with the comparator oral cladribine for consecutively included patients with active RMS. Randomization rituximab:cladribine is 1:1.
Who Masked: Outcomes Assessor
Masking Description: Two independent blinded radiologists assess the primary endpoint, New or enlarging T2 lesions. The blinding is asserted by transfer of deidentified MRIs to a Research server, from where the assessment is performed, so that the radiologists know only the ID, not the treatment allocation of the patients from whom the assess MRIs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Active Comparator): Biosimilar rituximab concentrate for solution for infusion
  Interventions: Biological: Rituximab
- Cladribine (Active Comparator): Mavenclad oral cladribine tablets
  Interventions: Drug: Cladribine

INTERVENTIONS:
Biological: Rituximab — Biosimilar rituximab concentrate for solution for infusion
  Arms: Rituximab
Drug: Cladribine — Mavenclad oral cladribine tablets
  Other Names: Mavenclad
  Arms: Cladribine

SUMMARY:
The main aim and overall objective of the study is to assess whether rituximab is non-inferior to cladribine for the treatment of relapsing MS. Secondly, the investigators will test specific blood and MRI biomarkers that may contribute to future personalized treatment for MS patients. Furthermore, the investigators want to evaluate the health economic consequences of the two therapies.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a demyelinating and neurodegenerative inflammatory disease of the central nervous system, affecting more than 12 000 patients in Norway and more than 2.2 mill patients worldwide.

Oral cladribine is one of the first choices for highly efficient disease modulatory treatment (DMT), while Rituximab is used off-label as DMT in relapsing MS. Large observational studies indicate good tolerance and treatment effect of rituximab in MS and studies from other diseases indicate a good safety profile. However, no phase 3 studies have been performed to test whether rituximab is as efficient as established MS treatments. Formal safety data is also lacking for the treatment with rituximab in MS.

The investigators will perform a prospective randomized open-label blinded endpoint multicenter non-inferiority study. The primary objective is to test whether rituximab is non-inferior to oral cladribine in the treatment of relapsing MS. 264 MS patients aged 18-65 years with relapsing MS will be recruited from 10 centers and followed for 96 weeks. The primary endpoint is difference in new T2 lesions between the groups. Furthermore, the investigators will test novel blood sample and MRI biomarkers to provide tools for personalized MS treatments. Finally, the health economic consequences of these treatment options will be evaluated.

This study will guide clinicians and patients in the future treatment choice for MS and can potentially make a huge impact on the costs of future MS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* A diagnosis of relapsing MS according to the 2017 McDonald criteria
* Disease activity seen as either a clinical relapse or MRI activity during the last 12 months
* EDSS between 0 and 5.5
* Thrombocytes and leukocytes within normal range, and lymphocytes above 0.8 x10 9/L before first dose of study medication
* A) For women of childbearing potential: accepting to use adequate contraception in the trial period. If randomized to cladribine, women who use systemic hormonal contraception must accept to use additional barrier contraception during each treatment cycle and for four weeks after each treatment cycle.
* B) For men: If randomized to cladribine, accepting to use adequate contraception in the safety period of 6 months after each treatment cycle.
* Able to understand written and spoken Norwegian or English
* Able to complete treatment or follow-ups in the study (e.g. no contraindications for MRI, severe psychiatric disease, drug abuse or plans of moving)
* Signed informed consent

Exclusion Criteria:

* Any contraindication or increased risk of side-effects from rituximab or cladribine (such as ongoing acute or chronic infection, live vaccination less than 4 weeks before start of treatment or planned live vaccination, immunocompromised, previous or active malignant disease, ongoing glucocorticoid treatment or allergy against any products of the medication)
* Previous use of any of cladribine, rituximab, alemtuzumab, ocrelizumab, hematopoietic stem cell therapy (HSCT) or other immunosuppression with long lasting effects
* Fingolimod or natalizumab treatment within the last six months before inclusion
* Current pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of new or enlarging cerebral MRI T2 lesions | Week 12-96
  The primary outcome is the number of new or enlarging cerebral MRI T2 lesions per patient from week 12 to week 96

SECONDARY OUTCOMES:
T2 lesions after 48 weeks | Week 12-48
  Number of new or enlarging cerebral MRI T2 lesions per patient from week 12 to week 48
Annual clinical relapse rate (ARR) | Week -2 to 96
  Annual clinical relapse rate (ARR) at 24, 48 and 96 weeks
Relapse-free patients | Week -2 to 96
  Proportion of relapse-free patients at 24, 48 and 96 weeks
Disability progression | Week -2 to 96
  Proportion of patients with 24 weeks confirmed disability progression (24-CDP) on EDSS at 48 and 96 weeks
Change in disability | Week -2 to 96
  Change in disability on the Expanded Disability Status Scale (EDSS) from week -2 to 48 and 96 weeks. Disability progression is defined as an increase in EDSS of at least 1.5 points if baseline EDSS was 0, 1 point with baseline EDSS 0.5-4.5 and 0.5 point with baseline EDSS 5-5.5. EDSS is a scale from 0-10 measuring neurological disability.

OTHER OUTCOMES:
MRI from baseline | Week -6 - 96
  Number of new or enlarging cerebral MRI T2 lesions from week -6 to week 12, 48 and 96
No evidence of disease activity (NEDA 3) | Week -2 - 96
  NEDA 3 (no evidence of disease activity) defined as no new or enlarging T2 lesions, no clinical relapse and no confirmed disability progression on EDSS from before treatment in week -2 to 48 and 96 weeks. Rate of NEDA in the two treatment groups are compared.
MRI contrast enhancing lesions | Week 12-96
  Number of new or persisting contrast enhancing (CE) MRI T1 lesions at 12, 48 and 96 weeks compared to previous scan
Patient reported outcome measures (PROMS) concerning work capacity | Week -2 - 96
  Patient self-evaluation with PROMS at week
  -2, 48 and 96 using questions about work capacity. The numerical values of the respones to the questions concerning adherence to work (percentage in full time work) in the two treatment groups are compared.
Patient reported outcome measures (PROMS) of fatigue | Week -2 - 96
  Patient self-evaluation with PROMS at week
  -2, 48 and 96 using questions about fatigue, the Fatigue Scale for Motor and Cognitive Functions (FSMC). The FSMC includes a Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') and produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue).The numerical values of the scores of the questionnaire in the two treatment groups are compared.
Patient reported outcome measures (PROMS) of anxiety and depression | Week -2 - 96
  Patient self-evaluation with PROMS at week
  -2, 48 and 96 using questions concerning anxiety and depression, Hospital Anxiety and Depression Scale (HADS). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.Thus minimum value is 0 (no anxiety or depression at all) and maximum value is 21 (severest grade of anxiety or depression).The numerical values of the scores of the questionnaire in the two treatment groups are compared.
Patient reported outcome measures (PROMS) of Health related quality of life | Week -2 - 96
  Patient self-evaluation with PROMS at week
  -2, 48 and 96 using questions concerning Health Related Quality of Life using the questionnaire EuroQol 5 Dimension scale (EQ5D). The respondents are asked to choose one of five statements which best describes their health status. Rated level can be coded as a number between 1-5, which indicates having no problems for 1, having slight problems for 2, having moderate problems for 3, having severe problems for 4, and having extreme problems for 5.The numerical values of the scores of the questionnaires in the two treatment groups are compared.
Patient reported outcome measures (PROMS) of treatment satisfaction | Week -2 - 96
  Patient self-evaluation with PROMS at week 48 and 96 using questions concerning treatment satisfaction, measured with the Treatment Satisfaction Questionnaire for Medicine (TSQM 1.4). The TSQM consists of fourteen questions distributed across four domains: effectiveness, side effects, convenience and global satisfaction. The score ranges from 0 to 100 in each domain and, the higher the score, the greater the patient satisfaction with medication. The numerical values of the scores of the questionnaires in the two treatment groups are compared.
Treatment adherence | Week 48-96
  Proportion of patients not receiving treatment per protocol at week 48 and 96
Safety endpoints blood sample: Occurrence of leukopenia indicated from blood samples | Week 0-96
  Occurrence of leukopenia grade 1 or 2 (mild), 3 or 4 (severe), according to World Health Organization (WH) using indicated from blood samples between first treatment at week 0 and end of study at week 96
Safety endpoints blood sample: Occurrence of lymphopenia indicated from blood samples | Week 0-96
  Occurrence of lymphopenia grade 1 or 2 (mild), 3 or 4 (severe), according to World Health Organization (WH) using indicated from blood samples between first treatment at week 0 and end of study at week 96
Safety endpoints blood sample: Occurrence of thrombocytopenia indicated from blood samples | Week 0-96
  Occurrence of thrombocytopenia grade 1 or 2 (mild), 3 or 4 (severe), according to World Health Organization (WH) using indicated from blood samples between first treatment at week 0 and end of study at week 96
Safety endpoints blood sample: Occurrence of anemia indicated from blood samples | Week 0-96
  Occurrence of anemia grade 1 or 2 (mild), 3 or 4 (severe), according to World Health Organization (WH) using indicated from blood samples between first treatment at week 0 and end of study at week 96
Safety endpoints adverse events | Week 0-96
  Adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR) reported between first treatment at week 0 and end of study at week 96
Blood sample neurofilament | Week -1 - 96
  Concentration of blood serum levels of neurofilament (NfL) at week -1, 51 and 96 weeks in the two treatment Groups are compared.
Blood sample glial fibrillary acidic protein | Week -1 - 96
  Concentration of blood serum levels of glial fibrillary acidic protein (GFAP) at week -1, 51 and 96 weeks in the two treatment Groups are compared.
Blood sample immunization antibodies for pneumococcus | Week -2 - 96
  Specific antibody titers for pneumococcus at week -2, 8, 51 and 96 are compared in the treatment Groups after immunization
Blood sample rituximab | Week -2 - 96
  Levels of rituximab in serum at week 8, 51 and 96 is related to MRI, relapse rate and EDSS in the rituximab treatment group
Blood sample rituximab antibody | Week -2 - 96
  Specific antibody titers at week 8, 51 and 96 of rituximab antibodies are correlated With rituximab concentration, MRI, EDSS and relapse rate in the rituximab treatment group
T2 lesion volume | Week 12-96
  T2 lesion volume at 12, 48 and 96 weeks are compared between the treatment groups
Brain volumes | Week 12-96
  Brain volumes at 12, 48 and 96 weeks are compared between the treatment groups
Advanced MRI analysis machine learning | Week 12-96
  Estimation of "Brain Age" at 12, 48 and 96 weeks Results of MRI analyses with and without AI and/or machine learning
Health economic analysis | -2 - 96
  Direct and indirect treatment costs (medication, out-patient clinic visits, hospitalizations related to treatment), working status) and health related quality of life (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Flistad Harbo, MD, PhD, Study Chair — Oslo University Hospital; Gro Owren Nygaard, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (11):
- Norway (11):
  - Department of Neurology - Drammen, Vestre Viken HF, Drammen, Buskerud
  - Department of Neurology - Lillehammer, SI Lillehammer, Lillehammer, Oppland
  - Department of Neurology, Stavanger universitetssykehus, Stavanger, Rogaland
  - Department of Neurology - Førde, Helse Førde HF, Førde, Sogn Og Fjordane
  - Department of Neurology - Skien, Sykehuset Telemark, Skien, Telemark
  - Department of Neurology - Tromsø, University Hospital of North Norway, Tromsø, Troms
  - Department of Neurology - Kristiansand, Sørlandet sykehus HF, Kristiansand, Vest-Agder
  - Department of Neurology - Tønsberg, Sykehuset i Vestfold HF, Tønsberg, Vestfold
  - Department of Neurology, Oslo University Hospital, Oslo
  - St. Olavs Hospital, Trondheim University Hospital, Trondheim
  - Department of Neurology - Kalnes, Sykehuset Østfold HF, Sarpsborg, Østfold fylke